CLINICAL TRIAL: NCT06105398
Title: Investigation Of The Effect Of Core Stability On Hand Functions In Patients Undergoing Rotator Cuff Surgery
Brief Title: the Effect of Core Stability on Hand Functions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gülçe İrem Yalçınkaya (Other)
Responsible Party: Sponsor-Investigator, Gülçe İrem Yalçınkaya, Principal Investigator, Pamukkale University
Organization: Pamukkale University (Other)
Other Study IDs: Pamukkale Universty
Record Dates: First submitted 2023-08-07; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Rotator Cuff Tear Arthropathy
Keywords: Hand Function, Core Stability
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients between the ages of 40-75 who had rotator cuff repair at least one year ago at the Orthopedics and Traumatology Clinic of Pamukkale University
  Interventions: Other: clinical evaluation
- Control group: healthy adults between the ages of 40-75
  Interventions: Other: clinical evaluation

INTERVENTIONS:
Other: clinical evaluation — clinical evaluation tests

SUMMARY:
Determining the factors affecting hand function after upper limb injuries is very important for maintaining independence in daily living activities. The aim of this study is to determine the relationship between core stability and hand function in patients undergoing rotator cuff surgery and to compare the results with healthy patients of a similar age. The aim of this study is to determine the relationship between core stability and hand function in patients undergoing artroscopic cuff surgery.

DETAILED DESCRIPTION:
The shoulder joint is a joint that is open to injuries due to its wide December of movement. For this reason, it is the most important cause of upper extremity pain.The most common cause of shoulder pain is rotator cuff injuries.Rotator cuff injuries are a painful problem of the shoulder that causes movement restriction, pain and impaired functional activities. Excessive use of the shoulder occurs as a result of impaired shoulder stability, November, muscle weakness, trauma. Although the prevalence of rotator cuff ruptures increases with age, they usually start at the age of 40 and the incidence increases by 54% at the age of 60 and by 60- 80% at the age of 80. It has a prevalence ranging from 20-50% in the general population. Arthroscopic repair has found widespread use due to the reasons that the protection of the adhesion site of the deltoid November, the diagnosis and treatment of concomitant intra-articular pathologies are easier, adhesions are less common, pain is less and rehabilitation after repair is easier.Core stability is considered very important in terms of biomechanical efficiency because it optimizes force production in all kinds of physical activities, from running to throwing, and minimizes the loads placed on the joints. However, there is little clarity about exactly what the anatomical and physiological characteristics of the structures that make up core stability are. However, core stability is defined as the ability to control the position and movement of the trunk on the pelvis to allow optimal production, transfer and control of force and movement to the terminal segment during activities. Core November muscle activity is best understood as the pre-programmed integration of regional, single-jointed and multi-jointed muscles to provide stability and November muscle activity is best understood as the pre-programmed integration of regional, single-jointed and multi-jointed muscles to produce movement. This results in the creation of proximal stability for distal mobility, a proximal-to-distal model of force generation, and interactive moments that move and protect the distal joints . Strong core stabilization minimizes the load on the vertebral column, increases the durability of the peripheral joints and also provides energy transfer to the distal segments. The relationship between core stability and limb Deceleration performance has been studied in athletes in general. However, most of the studies have focused on core stability and lower limb relationship.Evaluation of hand function and performance is important in terms of determining the person's skill level in daily life activities and demonstrating the effectiveness of rehabilitation.Hand function can be defined as the capacity of the hand for daily activities in connection with anatomical integrity, mobility, strength, sensation, coordination, age, gender, mental status, illness or trauma, and the condition of other proximal limb joints (shoulder, elbow, wrist). In order to determine which approaches are more effective in correcting the loss of function that occurs after various injuries and diseases, it is first necessary to have a good understanding of the factors that affect this performance.

ELIGIBILITY:
Inclusion Criteria:

* - Patients who have had rotator cuff repair done (at least one year ago)
* Non-rerupturants
* Those who have not suffered any other upper limb injuries after surgery
* Those who do not have any chronic diseases that can negatively affect ligament healing
* Those who do not have any spinal and lumbar region pathology
* Those who do not have lower back and back pain
* Those who do not have any neuromuscular diseases
* Those who can be cooperated

Exclusion Criteria For Volunteers:

* Patients who have not had rotator cuff repair
* Those who are recurrent
* Those who have suffered any other upper limb injury after surgery
* Those with any chronic diseases that can negatively affect ligament healing
* Those with any spinal and lumbar region pathology
* Those with lower back and back pain
* Those who have undergone spinal surgery
* Those with any neuromuscular disease
* Those who cannot establish coperation

Exclusion Criteria:

* Patients who did not complete the evaluations and wanted to leave voluntarily were excluded from the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study group: 47 patients between the ages of 40-75 Control group : 47 healthy adults between the ages of 40-75
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
hand dominance test | 1 year
  Edinburgh Hand Preference Survey
muscle strength test | 1 year
  Jamar Hand Dynamometer
Evaluation of reaction time test | 1 year
  Nelson hand reaction test
upper extremity function test | 1 year
  Q-DASH Survey
hand function test | 1 year
  Jebsen Taylor Hand Function Test
upper extremity balance test | 1 year
  Upper Extremity Y Balance Test
core stabilization test | 1 year
  Core Stabilization Assessment (trunk flexor, trunk extensor endurance, side plank, double straight leg lowering)
Pain scale | 1 year
  Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No